CLINICAL TRIAL: NCT05600166
Title: A Prospective Cohort Study Evaluating the Efficacy of a Double-layer Artificial Dermal Repair Material Combined With Growth Factors for Exposed Tendon Wounds
Brief Title: Double-layer Artificial Dermal Repair Material Combined With Growth Factors is Used for Exposed Tendon Wounds
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wang xingang (Other)
Responsible Party: Sponsor-Investigator, Wang xingang, Deputy Director, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: wxg1018
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Open Wound of Hip With Tendon Involvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Participants were treated with artificial dermal repair materials in combination with growth factors.
- Control group: Cases treated with a double layer of artificial dermal repair material

SUMMARY:
Compared with the combination of double-layer artificial dermal repair materials combined with growth factors, and the treatment methods using double-layer artificial dermal repair materials, the time and effect of the two treatment regimens on the function and appearance of wound repair with exposed tendon were different, as well as the medical costs.

DETAILED DESCRIPTION:
This study used a prospective cohort study to select all patients who met the inclusion criteria in six hospitals within six months after the start of the trial, including no less than 55 patients receiving artificial dermis combined with growth factor and no less than 110 patients receiving simple artificial dermal treatment, and the cumulative number of patients was not less than 110 patients, to compare the time and effect of the two treatment options on the functional and cosmetic restoration of upper limb wound repair with exposed tendons.

ELIGIBILITY:
Inclusion Criteria:

1. Elbow joint to fingertip area, soft tissue defect accompanied by tendon exposed fresh wound, tendon exposed wound area of 2~20cm2, wound area 5-600cm2, need to transplant autologous skin;
2. Incomplete aponeurosis;
3. Voluntarily sign the informed consent form. For persons with no or limited capacity for civil conduct, obtain the consent of their guardians and sign an informed consent form.

Exclusion Criteria:

1. Wound infection or suspected osteomyelitis;
2. Chronic wounds;
3. More than 2/3 of the exposed tendons are suspended on the wound surface;
4. Those with serious primary diseases such as cardiovascular and cerebrovascular, liver and kidney and hematopoietic system, which cannot be treated by surgery;
5. Those who are allergic to collagen and chondroitin sulfate;
6. Other persons that the investigator deems unsuitable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who met the inclusion criteria were selected for treatment at 6 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Wound closure evaluation | Two successive observations confirm the time when the wound is completely closed
  After transplantation of the autologous epidermis, it takes for the exposed tendon wound to heal 100%.
Wound closure evaluation | 7 days after the patient implanted the autologous blade thick skin tablet
  One week after transplantation of the autologous epidermis, the survival rate of skin grafting on the exposed tendon wound is localized.
Functional evaluation | 3 months after surgery
  Quick DASH
Functional evaluation | 6 months after surgery
  Quick DASH
Functional evaluation | 3 months after surgery
  Range of motion
Functional evaluation | 6 months after surgery
  Range of motion
Appearance evaluation | 3 months after surgery
  VSS（Vancouver scar scale） score of the receiving area .About scars, color 0~3 points; Thickness 0~4 minutes; Vascular distribution 0~3 points; Softness: 0~5 points. All the points are added together, the smaller the better.
Appearance evaluation | 6 months after surgery
  VSS（Vancouver scar scale） score of the receiving area .About scars, color 0~3 points; Thickness 0~4 minutes; Vascular distribution 0~3 points; Softness: 0~5 points. All the points are added together, the smaller the better.
Appearance evaluation | 3 months after surgery
  VSS（Vancouver scar scale） score of the the supply area.About scars, color 0~3 points; Thickness 0~4 minutes; Vascular distribution 0~3 points; Softness: 0~5 points. All the points are added together, the smaller the better.
Appearance evaluation | 6 months after surgery
  VSS（Vancouver scar scale） score of the supply area.About scars, color 0~3 points; Thickness 0~4 minutes; Vascular distribution 0~3 points; Softness: 0~5 points. All the points are added together, the smaller the better.